CLINICAL TRIAL: NCT00052481
Title: Health-Related Quality Of Life In Patients With Low Risk, Localized Prostate Cancer Randomized To Radical Prostatectomy Or Brachytherapy
Brief Title: Quality of Life in Patients Undergoing Surgery or Brachytherapy for Stage II Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACOSOG-Z0071; ACOSOG-Z0071; CDR0000258478 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of life questionnaire: Patients are randomized to 1 of 2 arms on ACOSOG-Z0070 (radical prostatectomy vs brachytherapy).
  Patients in both arms complete a quality of life questionnaire at baseline, 2 and 6 months after treatment, and then at 1, 2, 4, 7, and 10 years after treatment as part of ACOSOG-Z0071.
  Interventions: Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Quality of life assessment in patients undergoing prostate cancer treatment may help determine the intermediate-term and long-term effects of surgery and brachytherapy.

PURPOSE: Randomized clinical trial to study quality of life in patients undergoing radical prostatectomy or brachytherapy for stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare changes in health-related quality of life (HRQOL) in patients with stage II prostate cancer up to 2 years after treatment with radical prostatectomy or brachytherapy.
* Compare the effect of baseline HRQOL, age, and other covariates on HRQOL improvement or deterioration in these patients up to 10 years after these treatments.
* Compare the effect of treatment modality on HRQOL improvement or deterioration in these patients up to 10 years after these treatments.
* Compare the effects of treatment failure on HRQOL, in terms of disease progression, in these patients.

OUTLINE: Patients are randomized to 1 of 2 arms on ACOSOG-Z0070 (radical prostatectomy vs brachytherapy).

Patients in both arms complete a quality of life questionnaire at baseline, 2 and 6 months after treatment, and then at 1, 2, 4, 7, and 10 years after treatment.

PROJECTED ACCRUAL: A total of 500 patients (250 per group) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate within the past 120 days

  * Stage II disease (T1c-T2a, N0, M0)
* Concurrent enrollment on ACOSOG-Z0070

  * Not yet randomized to an intervention arm (radical prostatectomy or brachytherapy)
* Willing and able to complete heath-related quality of life questionnaires

PATIENT CHARACTERISTICS:

Age

* 75 and under

PRIOR CONCURRENT THERAPY:

Endocrine therapy

* More than 6 months since prior hormonal therapy for prostate cancer

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with adenocarcinoma of the prostate and previously enrolled on ACOSOG-Z0070.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2002-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
time to treatment failure | Up to 10 years

SECONDARY OUTCOMES:
disease progression | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandra G. Martin, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (13):
- United States (13):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington